CLINICAL TRIAL: NCT07396961
Title: Evaluation of the Consistency of the ASIS Line for Lumbar Level Identification in the Lateral Decubitus Position: Comparison With the Tuffier's Line
Brief Title: Consistency of ASIS Line vs. Tuffier's Line for Lumbar Level Identification
Status: Not yet recruiting | Type: Observational
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Sung Hyun Lee, Associate Professor, Kangbuk Samsung Hospital
Other Study IDs: 2026-01-002
Record Dates: First submitted 2026-01-30; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Spinal Anesthesia Evaluation; Lumbar Vertebrae
Keywords: vertebral level; Ultrasound; Tuffier's line; ASIS; Lateral decubitus position
MeSH Terms: interventions — Palpation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: Adult patients (aged 18-85) scheduled for spinal anesthesia or lumbar ultrasound
  Interventions: Diagnostic Test: Lumbar Ultrasound & Palpation

INTERVENTIONS:
Diagnostic Test: Lumbar Ultrasound & Palpation — Identification of vertebral levels using Tuffier's line (palpation) and ASIS line, followed by ultrasound verification.

SUMMARY:
Tuffier's line is commonly used as a landmark for estimating lumbar vertebral levels during spinal anesthesia. However, its accuracy can vary depending on factors such as age, sex, BMI, and posture. This study evaluates the consistency of an alternative landmark, the "ASIS line" (a line connecting both Anterior Superior Iliac Spines), for identifying lumbar levels in the lateral decubitus position. Researchers will mark both the ASIS line and Tuffier's line on participants and use ultrasound to verify the exact vertebral level where each line crosses the spine. The goal is to determine if the ASIS line provides a more consistent and reliable estimation of lumbar levels compared to Tuffier's line.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 85 years
* Patients scheduled for spinal anesthesia or lumbar ultrasound
* Participants who voluntarily agreed to participate and provided written informed consent

Exclusion Criteria:

* History of spinal surgery or spinal deformity
* Infection or wounds at the puncture site
* Inability to maintain the lateral decubitus position
* Congenital lumbosacral transitional vertebrae (e.g., sacralized L5 or lumbarized S1)
* Any other condition deemed unsuitable for the study by the investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting the study centers (Kangbuk Samsung Hospital or St. Vincent's Hospital) who are scheduled for spinal anesthesia or lumbar ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2027-02-20 (Estimated); Study Completion 2028-02-20 (Estimated)

PRIMARY OUTCOMES:
Consistency of Vertebral Level Identification (Standard Deviation) | Day 1 (Immediately during the ultrasound examination)
  The specific vertebral level where the ASIS line and Tuffier's line intersect the spine will be identified using ultrasound. The lumbar spine (from L2 upper to S1 upper) is divided into segments (e.g., L2=2, L3=3, L4=4, L5=5, S1=6). The consistency of each method is evaluated by calculating and comparing the standard deviation (SD) of the identified vertebral levels.

SECONDARY OUTCOMES:
Difference in Mean Intersection Level | Day 1
  Comparison of the mean vertebral levels identified by the ASIS line versus Tuffier's line to determine if there is a significant difference in the average level indicated.
Rate of Identification within L4-L5 Interspace | Day 1
  The percentage of cases where the identified line falls within the target L4-L5 interspace (or within ±1 interspace range).

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - St. Vincent's Hospital, Suwon, North Carolina
  - Kangbuk Samsung Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No